CLINICAL TRIAL: NCT06711471
Title: Phase II Study of Trifluridine/tipiracil (TAS-102), Bevacizumab, and Camrelizumab As a Third-line or Later-line Therapy for Patients with Metastatic Gastric Cancer
Brief Title: Trifluridine/tipiracil (TAS-102), Bevacizumab, and Camrelizumab As Third-line or Later-line Therapy of Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LIN YANG (Other)
Responsible Party: Sponsor-Investigator, LIN YANG, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4916
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer Adenocarcinoma Metastatic
MeSH Terms: interventions — Trifluridine; tipiracil; trifluridine tipiracil drug combination; Bevacizumab; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- trifluridine/tipiracil, bevacizumab, camrelizumab (Experimental): TAS-102 35mg/m² twice daily, orally on Days 1-5; Bevacizumab 5mg/kg intravenous infusion on Day 1; Camrelizumab 200mg intravenous infusion on Day 1; Repeat every 14 days.
  Interventions: Drug: trifluridine/tipiracil (TAS-102), bevacizumab plus camrelizumab

INTERVENTIONS:
Drug: trifluridine/tipiracil (TAS-102), bevacizumab plus camrelizumab — Patients enrolled in this study will receive trifluridine/tipiracil in combination with bevacizumab and camrelizumab, with a treatment cycle of 14 days, until disease progression, death, intolerable toxicity, or other criteria for discontinuation of study treatment as specified in the protocol (whichever occurs first).

SUMMARY:
For patients with metastatic gastric cancer, the efficacy of current standard treatments outlined in the guidelines is far from meeting the clinical demand. This study aims to explore the efficacy and safety of trifluridine/tipiracil (TAS-102), bevacizumab plus camrelizumab as a novel third-line or later-line therapy for metastatic gastric cancer patients.

DETAILED DESCRIPTION:
This study is an explorative prospective phase II clinical study. The study recruits patients with advanced gastric/gastroesophageal junction adenocarcinoma who have experienced disease progression after at least two lines of systemic therapy.

Participants must undergo screening tests within 28 days before treatment to determine their eligibility for the study. Patients who meet the inclusion criteria will receive treatment with trifluridine and tipiracil combined with bevacizumab and camrelizumab, with a treatment cycle of 14 days until disease progression, death, intolerable toxicity, or other criteria for terminating study treatment as specified in the protocol (whichever occurs first).

Tumor assessment will be conducted according to the RECIST 1.1 criteria. It will be performed by the researcher or designated research staff every 3 cycles after the start of treatment, until disease progression, death, the initiation of other anti-tumor treatments, or withdrawal of informed consent. Safety follow-up will be conducted after the last dose to monitor the resolution of adverse events. After treatment termination, participants will be followed up for survival every 90 days until death or loss of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histopathological confirmed gastric/GEJ adenocarcinoma.
2. The clinical stage was IV, according to AJCC 8th edition.
3. Patients had received at least two systematic therapies.
4. Patients had received or not received immunotherapy.
5. The patients received or did not receive anti-VEFGR targeted therapy in the last treatment (e.g., Bevacizumab, Ramucirumab, anti-VEGFR TKIs, etc.).
6. Age ≥18.
7. ECOG physical status score is 0-2 without deterioration within 2 weeks before the first administration of the investigational drug.
8. Adequate organ function according to the following laboratory test values:

   1. Hemoglobin value ≥90g/L.
   2. White blood cell count ≥3.5*109/L.
   3. Absolute neutrophil count ≥1.5*109/L.
   4. Platelet count ≥100*109/L.
   5. Serum creatinine ≤ upper limit of normal (ULN) or creatinine clearance ≥60ml/min.
   6. Total serum bilirubin ≤1.5 upper normal limit (ULN).
   7. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5 upper limit of normal value (ULN).
9. With a full understanding of the study, each participant volunteered to participate in this study and signed the informed consent (ICF) with good compliance and follow-up.

Exclusion Criteria:

1. Histopathological types other than adenocarcinoma include squamous cell carcinoma, adenosquamous carcinoma, neuroendocrine carcinoma, etc.
2. Known hypersensitivity or previous treatment with trifluridine/tipiracil or any of its components or excipients.
3. Known hypersensitivity to any component or excipients of bevacizumab.
4. Requirement for systemic corticosteroids (>10mg/day of prednisone or equivalent other corticosteroids, for a continuous treatment of ≥7 days) or immunosuppressive therapy within 14 days before enrollment; excluding inhaled or topical steroid use, or hormone therapy for adrenal insufficiency at physiological replacement doses; short-term (≤7 days) corticosteroids are allowed for prevention (e.g., contrast agent allergy) or treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity caused by contact allergens).
5. Receipt of a live vaccine (including attenuated live vaccines) or systemic immunostimulants (including but not limited to interferon or interleukin-2) within 28 days before enrollment.
6. Past or current interstitial pneumonia disease, except for those non-active and not requiring hormone therapy determined by the investigator.
7. Past or current autoimmune disease, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener's syndrome (granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophyseal inflammation, uveitis, autoimmune hepatitis, systemic sclerosis (scleroderma, etc.), Hashimoto's thyroiditis, autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome), etc. except for type I diabetes, hormonally replaced euthyroidism (including autoimmune thyroid disease causing hypothyroidism), psoriasis or vitiligo not requiring systemic treatment.
8. History of hypersensitivity, severe allergic reactions, or intolerance to antibody medications; history of significant allergies to drugs, foods, or other substances (e.g., severe allergic reactions, immunologically mediated hepatotoxicity, immunologically mediated thrombocytopenia, or anemia).
9. History of allogeneic bone marrow or organ transplantation.
10. Inability to swallow, intestinal obstruction, or other factors affecting drug intake and absorption.
11. Recurrent bleeding that cannot be controlled (as judged by the investigator to be at risk for major gastrointestinal bleeding, etc.).
12. Major surgery was performed within 4 weeks before the first study drug treatment (biopsy procedures excepted).
13. Concurrent malignancy within the past 5 years, except for those adequately treated cervical carcinoma in situ, localized squamous cell carcinoma of the skin, basal cell carcinoma, asymptomatic prostate cancer, ductal carcinoma in situ of the breast, well-differentiated thyroid cancer, or urinary tract epithelial cancer < T1, adequately treated lung carcinoma in situ, or other malignancies considered cured.
14. History of gastrointestinal perforation and/or fistula within the past 6 months, history of intestinal obstruction (including incomplete obstruction requiring parenteral nutrition), inflammatory bowel disease, or extensive bowel resection (partial colectomy or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
15. Any severe cardiac insufficiency, including left ventricular ejection fraction (LVEF) < 50%, congestive heart failure (CHF) ≥ grade 2 (CTCAE v5.0 or New York Heart Association grade ≥ 2), myocardial infarction, severe/unstable angina, stroke, or transient ischemic attack (TIA) within 6 months before enrollment.
16. Uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg) and diabetes (fasting blood glucose > 8.9 mmol/l).
17. History of ventricular tachycardia or torsades de pointes. Any resting ECG with significant clinical abnormalities in rhythm, conduction, or morphology, such as QTc > 450 msec for males, QTc > 470 msec for females, complete left bundle branch block, or third-degree atrioventricular block.
18. Active hepatitis B (must meet both HBsAg positive and HBV DNA ≥ 2000 IU/ml, or ≥ 104 copies, excluding hepatitis due to drugs or other causes), active hepatitis C (must meet both anti-HCV antibody positive and HCV RNA positive), syphilis (further testing for syphilis titer is required for those with positive syphilis antibodies), or human immunodeficiency virus (HIV) infection.
19. Pulmonary embolism or deep vein thrombosis occurring within 3 months before the first administration of the study drug (excluding thrombosis caused by catheters such as port, PICC, etc.).
20. Active pulmonary tuberculosis (TB), currently receiving anti-tuberculosis treatment, or those who have received anti-tuberculosis treatment within 1 year before the first dose.
21. Severe primary pulmonary disease, currently requiring continuous oxygen therapy for clinical active interstitial lung disease (ILD) or a history of pneumonia.
22. Uncontrolled active bacterial, viral, fungal, rickettsial, or parasitic infection requiring intravenous anti-infective treatment within 2 weeks before the first administration of the study drug.
23. Known history of substance abuse or drug addiction.
24. Pregnant or lactating women.
25. Fertile but unwilling to use effective contraceptive measures.
26. Any other diseases, metabolic disorders, or laboratory test abnormalities that the investigator has reason to suspect would make the patient unsuitable for treatment with the study drug, would affect the interpretation of the study results, or would place the patient at high risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-11-13 (Estimated); Study Completion 2027-11-13 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
12-week PFS rate | 12 weeks after the last patient was enrolled
6-month PFS rate | 6 months after the last patient was enrolled.
Disease Control Rate (DCR) | 2 years
Overall Survival (OS) | 2 years
Treatment-Related Adverse Events (TRAEs) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No